CLINICAL TRIAL: NCT07368790
Title: A Comparison of Postoperative Morphine Consumption in Patients Undergoing Elective Total Abdominal Hysterectomy With Preoperative Analgesia Intravenous Paracetamol Versus Placebo
Brief Title: Elective Total Abdominal Hysterectomy With Preoperative Analgesia Intravenous Paracetamol Versus Placebo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Savang Vadhana Memorial Hospital, Thailand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 011/2567
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Pain
Keywords: Paracetamol, Morphine, Total abdominal hysterectomy
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol (Experimental): Patients which recieved intravenous paracetamol preoperatively
  Interventions: Drug: Paracetamol
- Placebo (Placebo Comparator): Patients which recieved placebo preoperatively
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paracetamol — Patients receive IV paracetamol 1 gm Postoperatively morphine 0.1 mg/kg was given intravenous provided on demand at at 1, 6, 12, and 24 hours.
  Arms: Paracetamol
Drug: Placebo — Pateint recieved IV normal saline Postoperatively, pain was assessed intermittently using the NRS (์numeric rating scale) at 1, 6, 12, and 24 hours
  Arms: Placebo

SUMMARY:
The study aim to study to evaluate whether IV paracetamol reduces morphine use after TAH. Primary objective was to compare postoperative morphine consumption between the IV paracetamol and control groups.

and Secondary objective was to compare postoperative pain scores using the Numeric Rating Scale OR NRS

DETAILED DESCRIPTION:
We conducted a randomized, double-blind, placebo-controlled trial at our hospital (QSMH) , including women undergoing elective TAH The trial was conducted between October 2024 (two thousand twenty-four) and May 2025 (two thousand twenty-five) , with approval from the institutional review board.

Participants were randomized 1:1 (one to one) to receive IV paracetamol 1 g or IV normal saline, administered in the operating room before induction of anesthesia, Postoperatively, pain was assessed intermittently using the NRS (์numeric rating scale) at 1, 6, 12, and 24 hours, with morphine 0.1 mg/kg (zero point one milligrams per kilogram) Intravenous provided on demand.

The primary outcome was the number of morphine injections within 24 hours; the secondary outcome was NRS pain scores.

ELIGIBILITY:
Inclusion criteria

1. Female patients aged 30-50 years.
2. Scheduled to undergo total abdominal hysterectomy (TAH) at Queen Savang Vadhana Memorial Hospital at Sriracha
3. No history of allergy to paracetamol (acetaminophen) or morphine.
4. Normal renal function: serum creatinine ≤ 1.2 mg/dL.
5. No severe or recurrent liver disease, and AST or ALT ≤ 3× the upper limit of normal.
6. Able to communicate in Thai, complete the questionnaire, and provide written informed consent (no restriction on race or nationality).

Exclusion criteria

1. Incomplete medical record.
2. Use of any analgesic medications within 24 hours preoperatively.
3. Receipt of any postoperative analgesic other than morphine during the first 24 hours after surgery.
4. Withdrawal from the study.
5. Adverse reaction after administration of the study drug.
6. Concomitant surgery involving other organs (e.g., ovary or lymph nodes).

Ages: 30 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2024-10-10 (Actual); Primary Completion 2025-05-20 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Compare postoperative morphine consumption between the IV paracetamol and control groups. | at 1, 6, 12, and 24 hours postoperation

SECONDARY OUTCOMES:
Compare postoperative pain scores using the Numeric Rating Scale OR NRS | at 1, 6, 12, and 24 hours postoperation

CONTACTS AND LOCATIONS:
Overall Officials: Panumat Phungtippimanchai, Principal Investigator — Queen Savang Vadhana Memorial Hospital, Thailand
Locations (1):
- Queen Savang Vadhana Memorial Hospital, Thai Red Cross Society, Jermjomphon street, Chonburi, 20110,, Chon Buri, Thailand

IPD SHARING:
Plan to Share IPD: Undecided
data was save in form of microsoft excel spreadsheet and SPSS file